CLINICAL TRIAL: NCT02599935
Title: Impact on Nutrition and Quality of Life of Patients With Heart Failure After a Nurse Intervention on Nutrition Improvement
Brief Title: Nutritional Improvement in Chronic Heart Failure Patients
Acronym: VAINICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luis Guerra (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Luis Guerra, Nurse, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI11/02428
Record Dates: First submitted 2015-10-28; First posted 2015-11-09 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-11

CONDITIONS: Heart Failure
Keywords: Nutritional status; MNA; GSA
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- educational intervention and supplements (Experimental): structured educational intervention and dietary supplements
  Interventions: Dietary Supplement: Hypercaloric beverages; Other: educational structured counseling
- usual interventions (Active Comparator): Usual treatment without nutritional supplements or structured assessment
  Interventions: Other: standard treatment

INTERVENTIONS:
Dietary Supplement: Hypercaloric beverages — Nutritional supplement: Hypercaloric beverages
  Arms: educational intervention and supplements
Other: standard treatment — No other than standard treatment
  Arms: usual interventions
Other: educational structured counseling — Nutritional counseling leaded to patient and caregivers
  Arms: educational intervention and supplements

SUMMARY:
To assess the effect over the nutritional status in patients who are malnourished with chronic heart failure, of an educational intervention and the provision of nutritional supplements. Randomized clinical trial with blind assessors. Unicentric. Follow up: 12 months

DETAILED DESCRIPTION:
Randomized clinical trial with blinded evaluators. (The evaluators will not know the group the patients are assigned. Blinded evaluators are no responsible for randomization and intervention once the patients have been randomized). Patients will be recruited from the cardiology inpatient unit of tertiary hospital, before discharge. Patients will be divided in two groups randomly:

In one arm will be held a double intervention:

* A structured educational intervention oriented to the patient and primary caregiver, with respect to dietary habits, highly energetic and healthy food, the frequency and manner of eating, exercise and programming breaks.
* supplementation with dietary supplements, distinguishing one type of product or another, depending on whether the subject to study: diabetes and or kidney failure.

In the other arm of the study was carried out regular interventions

ELIGIBILITY:
Inclusion Criteria:

* adult patients with the diagnosis of heart failure: who inadvertently lost at least 5% of their "dry weight" in the last six months and / or moderately or severely malnourished according to the GSA and / or at risk or malnourished according to Mini Nutritional Assessment.
* Willing to participate by accepting and signing an informed consent.
* On treatment with inhibitors of angiotensin converting enzyme (ACE) inhibitors and / or antagonists of angiotensin II receptors (ARBs) and / or beta blockers.

Exclusion Criteria:

* Concurrent active cancer diagnosed.
* Previous history Dementia or severe cognitive impairment.
* Participation in another clinical trial simultaneously.
* Social or health condition that makes the patient impossible to follow the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2011-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change on nutritional status measured with Global Subjective Assesment | At inclusion , months 3 and 9

SECONDARY OUTCOMES:
Change on quality of life of patients measured with Minnesota Living With Heart Failure Questionnaire, after an educational intervention and nutritional supplement | At inclusion , months 3 and 9
Change on meters walked in six minutes (functional capacity), after the intervention | At inclusion , months 3 and 9
Number of readmission. | at month 12

CONTACTS AND LOCATIONS:
Overall Officials: Luis Guerra, Nurse, Principal Investigator — Hospital General Universitario Gregorio Maranon
Locations (1):
- Servicio de Nefrología Hospital General universitario Gregorio Maranon, Madrid, Madrid, Spain